# Delving Into Participation Patterns in Social Anxiety Clinical Trials and Investigating Engagement Trends Among Individuals Impacted by the Disease

An Informed Consent For Patients With Social Anxiety in <a href="Power">Power</a> <a href="Clinical Trial's">Clinical Trial's</a> Observational Study

Date: August 25, 2023

**Understanding This Informed Consent Document** 

If you are presented with the task of completing this document, it signifies your potential inclusion in an observational clinical trial designed specifically for individuals dealing with social anxiety. This document functions as an encompassing guide, unveiling the study's overarching aims, intricate execution plan, and multifaceted implications, both positive and potentially otherwise. Thoroughly contemplating your possible participation before arriving at a decision holds paramount importance, and seeking advice from a trusted doctor can provide invaluable perspectives. If any elements of the information contained here seem unclear or if questions arise, be assured that the researcher is readily available to offer clarifications.

# Objective of the Investigation

Social anxiety, also known as social anxiety disorder, is a mental health condition characterized by an intense and persistent fear of social situations or interactions. People with social anxiety often experience significant distress and anxiety when faced with social gatherings, public speaking, meeting new people, or other situations that involve potential scrutiny or evaluation by others.

Individuals with social anxiety may have irrational fears of being judged, embarrassed, or humiliated in social settings. This fear can be so overwhelming that it leads to avoidance of certain situations altogether. The anxiety can manifest as physical symptoms like sweating, trembling, a rapid heart rate, nausea, and even panic attacks.

Clinical trials specifically addressing social anxiety play a pivotal role in assessing the safety and efficacy of novel treatments for this condition. These trials are crucial in determining whether emerging treatments surpass existing options and provide substantial evidence to support their wider implementation.

This study specifically focuses on exploring the experiences of individuals diagnosed with social anxiety as they actively participate in a unique clinical trial involving medical interventions. The primary emphasis centers on closely analyzing trial completion rates and instances of voluntary withdrawal among these participants.

#### Delving into the Heart of Observational Studies

By becoming a participant in this medical trial, you immerse yourself in an observational study, a unique facet of clinical research meticulously designed to gather insights through the unaltered observation of individuals while maintaining their care plans.

Researchers will solely engage in observing your journey, meticulously assessing the outcomes of your condition without introducing any changes. This particular trial design plays a pivotal role in enriching our comprehension of the inherent progression of a specific medical condition and its effects on those who bear its diagnosis. By actively engaging in this observational study, you become an active contributor to expanding the boundaries of medical knowledge and fostering improvements in the care extended to individuals grappling with the same affliction.

# Contrasting This Trial Against Other Social Anxiety Cancer Clinical Trials

Recognizing the distinctive nature of this clinical trial is paramount. It operates within an observational framework, implying that your involvement will not encompass the administration of specific treatments or interventions. However, it is essential to grasp the comprehensive spectrum of social anxiety clinical trials, which encompasses interventional studies that entail participants undergoing specific treatment regimens.

Crafting an informed decision regarding your potential participation in a clinical trial requires an active approach involving exploration and comparison among diverse studies. A wealth of information pertaining to <u>studies related to social anxiety</u> is accessible through platforms like clinicaltrials.gov. Additionally, Power's dedicated online platform provides a comprehensive compilation of ongoing <u>social anxiety clinical trials</u> actively seeking participants. Through diligent research and an in-depth understanding of varied clinical trial formats, you empower yourself to confidently shape your participation decision.

#### Active Involvement in Clinical Trial Surveys

Within the context of this observational clinical trial, we extend a sincere invitation for you to actively contribute your experiences. This venture entails your periodic completion of questionnaires every two weeks, a commitment estimated to require approximately 20-30 minutes of your valuable time. Furthermore, at quarterly intervals, we are fully prepared to arrange check-in calls, an arrangement that will persist as long as your engagement in the trial endures.

Emphasizing the utmost significance, it is important to note that your participation in the survey phase of the trial is entirely voluntary. The autonomy to decide whether to address specific questions or the entirety of the questionnaire rests entirely with you. Moreover, you retain the independence to conclude your participation in the trial whenever you deem fit. Recognizing that the decision to participate in a clinical trial is deeply personal, our unwavering commitment lies in providing the necessary support. Your privacy and comfort remain our steadfast priorities, and we are dedicated to respecting and supporting your decision-making journey throughout the unfolding of the trial.

# Safeguarding the Confidentiality of Your Answers

Preserving the highest level of confidentiality for your information remains an absolute priority throughout the duration of this clinical trial. To ensure your anonymity, we kindly request that you refrain from including any personal or identifiable details in your responses to the questionnaires. The dedicated research team is resolute in their commitment to enhancing the shield of your confidentiality. However, it's important to acknowledge that specific legal situations may arise, requiring the disclosure of your data.

#### Possible Dangers

Amid the commendable advancement propelled by clinical trials, it remains pivotal to recognize the potential health hazards that participants might encounter, especially in trials examining new treatments.

Nonetheless, our observational clinical trial charts a distinct path, actively countering these risks by sidestepping the incorporation of novel interventions for participants. Rather, our primary focus centers on meticulous observation and measuring outcomes, a strategy designed to prevent any unwarranted health risks from entering the equation.

#### **Projected Gains**

While immediate advantages might not be immediately evident for individuals partaking in this observational clinical trial, their engagement carries the potential to extend its influence to others. The wealth of data accumulated from participants will fuel the refinement of future strategies for enrolling social anxiety patients, potentially paving the way for expanded avenues of medical research. Through their participation in this clinical voyage, individuals have the capacity to act as catalysts for transformative change within the domain of medical research, potentially reshaping the course for upcoming social anxiety patients.

# Exploring the Depths of Inclusivity in Clinical Trials

For those who possess a deep curiosity to delve into the intricate realm of representation in clinical trials, a plethora of online resources eagerly await your active engagement.

Whether your aim is to decipher the intricacies of challenges and opportunities surrounding clinical trial diversity, or you simply aspire to enrich your personal understanding, these sources can serve as illuminating guides:

<u>DuMont, Mieke, Alyssa Agostinis, Kiran Singh, Evan Swan, Yvonne Buttle, and Daniela Tropea. "Sex representation in neurodegenerative and psychiatric disorders' preclinical and clinical studies." *Neurobiology of Disease* (2023): 106214.</u>

Van IJzendoorn, Marinus H., and Marian J. Bakermans-Kranenburg. "The distribution of adult attachment representations in clinical groups: A meta-analytic search for patterns of attachment in 105 AAI studies." (2008).

#### Confirmation of Informed Choice

I hereby confirm that I have dedicated considerable time to comprehensively grasp and internalize the content contained within the informed consent form, either through a self-guided examination or with the assistance of a trusted individual who has conveyed its essence to me. All queries and uncertainties that occupied my thoughts have been diligently addressed to my complete satisfaction.

I am fully aware that my participation in this study is a result of my voluntary decision, and I retain the exclusive right to withdraw my consent without any obligation to provide justification or assume financial responsibilities. It has been expressly communicated to me that a duplicate of this informed consent form will be provided for my personal records.

Having thoroughly contemplated and evaluated the entirety of the information presented to me, I hereby extend my concurrence to engage in this study, reflecting my independent and informed choice.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| <br>Date |

### Confirmation by Informed Consent Facilitator

I confirm with conviction that I have engaged in a comprehensive dialogue with the participant, systematically unveiling the intricacies encompassed within this written document. My objective was to ensure that the participant grasps the trial's overarching objectives, employed methodologies, potential risks and benefits, as well as other critical elements intrinsic to the clinical trial for social anxiety.

Adequate space was provided for the participant, fostering the emergence of questions and facilitating the clarification of uncertainties or misconceptions. It is of utmost importance to underline that the participant's engagement in this trial is an outcome of their voluntary decision, and they possess the absolute prerogative to discontinue their involvement at any juncture, driven by any rationale, without incurring any financial obligations.

Following the participant's provision of consent, a diligently preserved duplicate of this written document was handed to them, serving as a repository for their individual records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| Date |